CLINICAL TRIAL: NCT02112500
Title: A Pilot Study for the Efficacy and Safety of Mesenchymal Stem Cell in Acute Severe Respiratory Failure.
Brief Title: Mesenchymal Stem Cell in Patients With Acute Severe Respiratory Failure
Acronym: STELLAR
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Sang Bum Hong, MD, Professor of Ulsan University College of Medicine, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STELLAR-Pilot
Record Dates: First submitted 2014-03-30; First posted 2014-04-14 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2016-01

CONDITIONS: Respiratory Distress Syndrome, Adult
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mesenchymal Stem Cell Infusion (Experimental): Mesenchymal stem cells cultured and extracted from bone marrow of enrolled patients are infused.
  Interventions: Biological: Mesenchymal Stem Cell

INTERVENTIONS:
Biological: Mesenchymal Stem Cell — Mesenchymal stem cells will be intravenously infused. Mesenchymal stem cells will be cultured and extracted from the bone marrow of the patients.
  Other Names: Lungcellgram

SUMMARY:
Although the advent of advanced medical support for respiratory failure, the mortality rate of acute severe respiratory failure is still high and the life quality is frequently compromised from pulmonary fibrosis.

The investigators hypothesize that the treatment using mesenchymal stem cell can be beneficial in patients with respiratory failure. The present study is a pilot study evaluating the efficacy and safety of mesenchymal stem cell treatment in patients with respiratory failure.

DETAILED DESCRIPTION:
Although the advent of advanced medical support for respiratory failure, the mortality rate of acute severe respiratory failure is still reported to be more than 40%. The respiratory distress syndrome may develop in all ages resulting in progressive pulmonary fibrosis. A number of survivors from respiratory failure suffer from the sequelas of pulmonary fibrosis.

However, the treatments of respiratory failure are limited to the correction of baseline disease, cardiopulmonary support, and conservative management to minimize the lung injury. There has not been any effective and specific treatment for respirator distress nor medicine to reduce mortality.

There have been reports of mesenchymal stem cell experimental animals with chronic obstructive pulmonary disease, interstitial lung disease, and sepsis. In addition, the mesenchymal stem cell treatment showed beneficial effect in bleomycin endotoxin induced lung injury.

Authors hypothesize that the mesenchymal stem cell treatment in patients with respiratory failure will show efficacy. We would conduct the present pilot study to evaluate the efficacy and safety in patients with respiratory failure and intend to suggest an additional alternative treatment option for those without additional treatment option.

ELIGIBILITY:
Inclusion Criteria:

* Ventilator care from respiratory failure
* Ventilator care for 7 or more days
* at least one of the followings

  1. PaO2/FiO2 = 200 or less when PEEP 5 cmH2O or more.
  2. PaCO2 = 50 mmHg or more when plateau pressure of 30 cmH2O or more.
  3. pH = 7.25 or less when plateau pressure of 30 cmH2O or more.
  4. No other treatment option except for lung transplantation and not candidate for recipient (organ failure, comorbid infection, economy,...)
  5. Ventilatory care with weaning failure 3 times or more
  6. Ventilator care requiring 7 days or more from the first self respiration to weaning of ventilator.

     * PEEP, positive endexpiratory pressure

Exclusion Criteria:

* Severe aplastic anemia
* Malignant hematologic disorder or history of stem cell treatment.
* Currently uncontrolled malignancy or history of solid cancer within 2 years
* HIV Infection
* Expected life < 3 months from other cause than the respiratory failure
* Pregnancy or breast feeding
* Expected hypersensitivity for study drug

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-02; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Oxygen index at 3 days after mesenchymal stem cell infusion | 3 days after mesenchymal stem cell infusion
  Oxygen index at 3 days after mesenchymal stem cell infusion. Oxygen index is calculated as follows; ((FiO2) x (Mean airway pressure)) / (PaO2)

SECONDARY OUTCOMES:
Lung mechanics | at 3, 14, and 28 days after mesenchymal stem cell infusion
  Lung mechanics includes arterial oxygen saturation, tidal volume, minute ventilation, and ratio of PaO2/FiO2.
Hemodynamic parameters | at 3, 14, and 28 days after mesenchymal stem cell infusion
  Systolic, diastolic, and mean arterial blood pressure Amount of required vasopressor Heart rate
Mortality | at 14 and 28 days after mesenchymal stem cell infusion
  Death from any cause at 14 and 28 days after mesenchymal stem cell infusion
Plasma cytokines | at 3, 14, and 28 days after mesenchymal stem cell infusion
  Interleukin (IL)-1, IL-6, IL-8, and IL-10
Markers for inflammation and infection | at 3, 14, and 28 days after mesenchymal stem cell infusion
  Lactate, DIC score, SOFA score, C-reactive protein, and procalcitonin
Ventilator weaning parameters | at 3, 14, and 28 days after mesenchymal stem cell infusion
  Failure of ventilator weaning, weaning time, ventilation time
ICU and hospital stay | at 28 days after mesenchymal stem cell infusion
  Total duration of ICU stay and hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Sang Bum Hong, M.D., Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Background] Calfee CS, Matthay MA. Nonventilatory treatments for acute lung injury and ARDS. Chest. 2007 Mar;131(3):913-920. doi: 10.1378/chest.06-1743. PMID 17356114
- [Background] Rubenfeld GD, Caldwell E, Peabody E, Weaver J, Martin DP, Neff M, Stern EJ, Hudson LD. Incidence and outcomes of acute lung injury. N Engl J Med. 2005 Oct 20;353(16):1685-93. doi: 10.1056/NEJMoa050333. PMID 16236739
- [Background] D'Agostino B, Sullo N, Siniscalco D, De Angelis A, Rossi F. Mesenchymal stem cell therapy for the treatment of chronic obstructive pulmonary disease. Expert Opin Biol Ther. 2010 May;10(5):681-7. doi: 10.1517/14712591003610614. PMID 20384521
- [Background] Lee JW, Gupta N, Serikov V, Matthay MA. Potential application of mesenchymal stem cells in acute lung injury. Expert Opin Biol Ther. 2009 Oct;9(10):1259-70. doi: 10.1517/14712590903213651. PMID 19691441
- [Background] Stagg J. Immune regulation by mesenchymal stem cells: two sides to the coin. Tissue Antigens. 2007 Jan;69(1):1-9. doi: 10.1111/j.1399-0039.2006.00739.x. PMID 17212702
- [Background] Gupta N, Su X, Popov B, Lee JW, Serikov V, Matthay MA. Intrapulmonary delivery of bone marrow-derived mesenchymal stem cells improves survival and attenuates endotoxin-induced acute lung injury in mice. J Immunol. 2007 Aug 1;179(3):1855-63. doi: 10.4049/jimmunol.179.3.1855. PMID 17641052
- [Background] Lee JW, Fang X, Gupta N, Serikov V, Matthay MA. Allogeneic human mesenchymal stem cells for treatment of E. coli endotoxin-induced acute lung injury in the ex vivo perfused human lung. Proc Natl Acad Sci U S A. 2009 Sep 22;106(38):16357-62. doi: 10.1073/pnas.0907996106. Epub 2009 Aug 31. PMID 19721001
- [Background] Ortiz LA, Dutreil M, Fattman C, Pandey AC, Torres G, Go K, Phinney DG. Interleukin 1 receptor antagonist mediates the antiinflammatory and antifibrotic effect of mesenchymal stem cells during lung injury. Proc Natl Acad Sci U S A. 2007 Jun 26;104(26):11002-7. doi: 10.1073/pnas.0704421104. Epub 2007 Jun 14. PMID 17569781
- [Background] Moodley Y, Atienza D, Manuelpillai U, Samuel CS, Tchongue J, Ilancheran S, Boyd R, Trounson A. Human umbilical cord mesenchymal stem cells reduce fibrosis of bleomycin-induced lung injury. Am J Pathol. 2009 Jul;175(1):303-13. doi: 10.2353/ajpath.2009.080629. Epub 2009 Jun 4. PMID 19497992
- [Background] Rojas M, Xu J, Woods CR, Mora AL, Spears W, Roman J, Brigham KL. Bone marrow-derived mesenchymal stem cells in repair of the injured lung. Am J Respir Cell Mol Biol. 2005 Aug;33(2):145-52. doi: 10.1165/rcmb.2004-0330OC. Epub 2005 May 12. PMID 15891110
- [Background] Zhen G, Liu H, Gu N, Zhang H, Xu Y, Zhang Z. Mesenchymal stem cells transplantation protects against rat pulmonary emphysema. Front Biosci. 2008 May 1;13:3415-22. doi: 10.2741/2936. PMID 18508443